CLINICAL TRIAL: NCT05585944
Title: " Effect of Single-nucleotide Polymorphism of CD40 Gene rs1883832 C/T on the Risk of Immune Thrombocytopenic Purpura "
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nagwa Mohamed Aboelmahasen, assisstant lecturer of clinical and chemical pathology department, Sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-22-10-21
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Immune Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): healthy participants
  Interventions: Diagnostic Test: Genotyping of rs1883832C/T related single-nucleotide polymorphism
- cases (Active Comparator): cases of immune thrombocytopenic purpura
  Interventions: Diagnostic Test: Genotyping of rs1883832C/T related single-nucleotide polymorphism

INTERVENTIONS:
Diagnostic Test: Genotyping of rs1883832C/T related single-nucleotide polymorphism — Genotyping of rs1883832C/T related single-nucleotide polymorphism by real time pcr
  Other Names: ANA test.

SUMMARY:
Immune thrombocytopenia is an acquired autoimmune disease, in which platelets are opsonized by auto-antibodies and destroyed by phagocytic cells .Genetic polymorphisms in the immune mediators have been suggested to play a pivotal role in the pathogenesis of many autoimmune disorders . Several genetic polymorphisms of the immune system genes have been described in ITP such as interleukins, tumor necrosis factors (TNF) alpha and beta, and interferon-gamma., These polymorphisms were found to be associated with an increased risk of ITP progression or exacerbation .CD40 is a co-stimulatory 4348 kDa glycoprotein molecule composed of 277 amino acid residues which belongs to the tumor necrosis family. It is encoded by a gene which is located at chromosome 20q11-13, expressed mainly on antigen presenting cells (APCs), some non-immune cells and tumors.Antinuclear antibodies (ANA) is a collective term for a large and heterogeneous group of circulating autoantibody. Reflecting their clinical importance, ANA are diagnostic, prognostic or classification criteria for many autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* sign an informed written consent from the patients or their parents
* patient with newly diagnosed ITP
* patient age > 1 year and < 65 years and both sexes are included.

Exclusion Criteria:

* Refusal to sign an informed written consent
* patient with persistent ITP, patient with secondary immune thrombocytopenia
* patient age < 1 year or > 65 years.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
rs1883832C/T related single-nucleotide polymorphism | 6 months
  effect of single-nucleotide polymorphism of CD40 gene (rs1883832 C/T) on the risk of immune thrombocytopenic purpura

SECONDARY OUTCOMES:
ANA | 6 months
  ANA in immune thrombocytopenic purpura

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Behzad MM, Asnafi AA, Jalalifar MA, Moghtadaei M, Jaseb K, Saki N. Cellular expression of CD markers in immune thrombocytopenic purpura: implications for prognosis. APMIS. 2018 Jun;126(6):523-532. doi: 10.1111/apm.12853. PMID 29924452
- [Background] Chen JM, Guo J, Wei CD, Wang CF, Luo HC, Wei YS, Lan Y. The association of CD40 polymorphisms with CD40 serum levels and risk of systemic lupus erythematosus. BMC Genet. 2015 Oct 16;16:121. doi: 10.1186/s12863-015-0279-8. PMID 26474561
- [Background] Favaloro EJ. How to Generate a More Accurate Laboratory-Based International Normalized Ratio: Solutions to Obtaining or Verifying the Mean Normal Prothrombin Time and International Sensitivity Index. Semin Thromb Hemost. 2019 Feb;45(1):10-21. doi: 10.1055/s-0038-1667342. Epub 2018 Aug 22. PMID 30134448
- [Background] Morodomi Y, Kanaji S, Won E, Ruggeri ZM, Kanaji T. Mechanisms of anti-GPIbalpha antibody-induced thrombocytopenia in mice. Blood. 2020 Jun 18;135(25):2292-2301. doi: 10.1182/blood.2019003770. PMID 32157300